CLINICAL TRIAL: NCT00346294
Title: An Open-Label Study to Assess the Rate of Failure of an Enbrel® (Etanercept) SureClick™ Auto-injector in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050207
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Device; Auto-injector; SureClick; Enbrel; Etanercept
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

ARMS (1):
- Single-Arm (Other): Open-lable Single Arm Study
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Intervention type was to study the drug delivery method.

SUMMARY:
An open-label, single arm study to estimate the rate of failure of the Enbrel® SureClick™ Auto-injector in RA subjects.

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of rheumatoid arthritis

* RA subjects
* 18 years or older
* Currently taking etanercept in pre-filled syringes for at least 4 weeks
* Subjects must give written informed consent
* Subjects must be able to read and write in English Exclusion Criteria: - Subject is not using adequate contraception
* Subject is pregnant or breast feeding
* Significant concurrent medical diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To estimate the rate of failure of the Enbrel® SureClick™ Auto-injector in RA subjects. | 22 Days

SECONDARY OUTCOMES:
To estimate the rate of failure of the Enbrel® SureClick™ Auto-injector at the subject level in RA subjects. | 22 Days
To determine the rate of failed drug deliveries (as opposed to device failures). | 22 Days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com